CLINICAL TRIAL: NCT03903744
Title: CardioneuROablation for Reflex Syncope: Effects on autonoMic cArdiac Regulation and Efficacy Assessment - the Roman Syncope Study.
Brief Title: Cardioneuroablation for Reflex Syncope
Acronym: ROMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Prof. Piotr Kulakowski, Principal Investigator, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113/PB/2018
Record Dates: First submitted 2019-03-30; First posted 2019-04-04 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Syncope, Vasovagal
Keywords: syncope; cardioneuroablation; cardioneuromodulation
MeSH Terms: conditions — Syncope, Vasovagal; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Patients treated with cardioneuroablation.
  Interventions: Procedure: Cardioneuroablation
- Control arm (Active Comparator): Patients treated with standard non-pharmacological methods.
  Interventions: Procedure: Cardioneuroablation

INTERVENTIONS:
Procedure: Cardioneuroablation — The electroanatomical map of the right (RA) and left (LA) atrium will be created and anatomically-based ablation of GP will be performed. Ablation in the RA is started from the supero-posterior area (superior right atrial GP), to the middle-posterior area (posterior right atrial GP). In the LA, ablation is started at the site of the anterior right GP and is continued downwards along the anterior part of a common vestibulum of the right pulmonary veins (PV), opposite to the right-sided ablation lesions. Finally, area of right inferior GP, close to the RIPV is ablated under intracardiac echocardiography control. Using this technique, GP's located close to the left PV are not ablated. We use a pure anatomic approach without identification of GP.
  Other Names: Cardioneuromodulation

SUMMARY:
Aim. To assess the effects of cardioneuroablation (CNA) on cardiac autonomic regulation and syncope recurrences in patients with vasovagal syncope (VVS), and to compare this novel approach with standard non-pharmacological treatment.

Measurements.

1. Before CNA:

   1. Detailed history taking and assessment of eligibility
   2. Baseline 12-lead ECG for heart rate assessment, morphology and duration of the P wave and PR interval
   3. 24-hour Holter ECG for heart rhythm (mean, minimal, maximal, pauses) and heart rate variability (HRV) assessment
   4. Passive tilt test (70 degrees, 45 minutes) to fulfill inclusion criterion and to assess baseline autonomic parameters such as HRV and baroreflex sensitivity (BRS) using sequential method. These parameters will be calculated from 5 min recordings before and after orthostatic stress (tilt).
   5. Atropine test - positive response to intravenous atropine in a dose of 2 mg defined as at least 30% increase in sinus rate compared with baseline value
   6. Assessment of quality of life using the SF-36 questionnaire
   7. Implantable Loop Recorder (ILR) implantation 2-3 days before CNA
2. During CNA:

   1. Heart rate before and immediately after CNA
   2. Episodes of bradycardia (sinus arrest or atrio-ventricular block) during application of RF to GP.
   3. Standard electrophysiological parameters (sinus node recovery time, corrected sinus recovery time, refractory atrio-ventricular node, atrio-ventricular conduction - Wenckebach point, A-H and H-V intervals) will be assessed before an immediately after CNA
   4. Atropine test (2 mg) will be repeated immediately after CNA.
3. After CNA:

   1. 1-2 days after CNA standard ECG
   2. Follow-up: 3, 12 and 24 months after CNA assessment of symptoms, 12 lead standard ECG, control of ILR, 24-hour Holter ECG, tilt test and atropine test will be performed. Additionally, quality of life will be assessed using SF-36 questionnaire

Anticipated results.

1. CNA performed with technique used in the present study is effective in > 90% of patients.
2. CNA-induced changes in analysed ECG and autonomic parameters predict CNA efficacy

DETAILED DESCRIPTION:
Introduction.

Reflex syncope due to vasovagal reaction is the most frequent cause of transient loss of consciousness (TLOC) in general population. [1-4] It markedly decreases quality of life and may lead to injury. [5, 6] The mechanism of vasovagal syncope (VVS) is complex. One of the most important mechanisms is enhanced parasympathetic activity triggered by abnormal mechanoreceptor reflex and other mechanisms. This leads to prolonged asystole and/or vasodilatation, resulting in syncope. [7] Treatment of VVS remains a challenge. Non-pharmacological treatment such as fluid and salt intake, avoiding situations triggering syncope or tilt training is not effective in a significant proportion of subjects with syncope. Pharmacotherapy is even less effective. Syncope recurs in 25-65% of patients. Alternative therapy, especially in patients with prolonged asystole, is pacemaker implantation, recommended by the guidelines in patients aged > 40 years with documented spontaneous cardioinhibitory VVS and severe symptoms. However, permanent pacing occurs ineffective in at least 25% of patients. In addition, VVS occurs predominantly in young persons in whom permanent pacing should be avoided as much as possible. [8-13] Thus, the need for new treatment options in VVS is clear.

Ablation for atrial fibrillation (AF) has been successfully performed for almost two decades. Apart from pulmonary vein isolation which is a corner stone of AF ablation, autonomic control of the heart is modified by ablation of ganglionated plexi (GP). It has been well documented that in some patients GP ablation increases the success rate of ablation, especially in patients with vagally-mediated AF. Thus, the technique of GP ablation, mainly using the radio-frequency energy, is well established and safe.

Based on data coming from GP ablation during AF procedures, this method has been recently proposed for patients with VVS. The postulated beneficial mechanisms of GP ablation in VVS are attenuation of parasympathetic activity, leading to elimination or reduction reflex asystole and bradycardia. To date, a few case series consisting of up to 70 patients demonstrated very promising results. [15-18]. However, this experience is limited to a few centers. Also, the optimal methodology of the procedure, called cardioneuroablation (CNA) or cardioneuromodulation, is not known. There is no consensus yet as to how many GP's, in both atria or only in the right atrium, in which order and to what extent should be ablated. Moreover, mechanisms responsible for beneficial effects of CNA as well as methods assessing it's efficacy are not clear.

Aim. To assess the effects of CNA on cardiac autonomic regulation and syncope recurrences in patients with VVS, and to compare this novel approach with standard non-pharmacological treatment.

Hypothesis. CNA using GP ablation causes significant changes in autonomic control of the heart, predominantly parasympathetic withdrawal, which is associated with long-term efficacy of the procedure, and is significantly more effective than standard non-pharmacological therapy.

Methods. This is an open-label, randomized, controlled, prospective study.

Study group. Forty consecutive patients with recurrent cardioinhibitory or mixed VVS will be included between August 2018 and July 2021.

The patients will be randomized into 2 groups:

1. Treatment arm (n=20): CNA
2. Control arm (n=20): standard non-pharmacological treatment The patients from the control arm will be allowed to cross over to the CNA group if syncopal episode occurs despite adherence to the non-pharmacological recommendations.

The number of 40 patients will be enough to demonstrate superiority of CNA over standard approach, assuming that the effectiveness of CNA will be over 90%, and the effectiveness of the standard non-pharmacological treatment will be 50%.

Inclusion criteria:

1. At least one documented spontaneous VVS during preceding 12 months or one syncope in history leading to injury and minimum 2 presyncopal events during preceding 12 months, refractory to all recommended types of standard treatment.
2. In case of lack of ECG documentation during spontaneous syncope and history suggesting reflex syncope, at least 3 seconds of asystole due to sinus arrest or atrio-ventricular block with syncope or bradycardia <40 beats per minute with syncope or presyncope during baseline tilt test
3. Sinus rhythm during ECG and tilt test
4. Significantly decreased quality of life due to syncope
5. Positive response to atropine test
6. Obtained written informed consent.

Exclusion criteria:

1. Other possible and treatable causes of syncope such as significant cardiac disease, cardiac arrhythmia or abnormalities of vertebro-basiliar arteries
2. History of stroke or TIA
3. History of cardiac surgery
4. Contraindications to ablation in the right or left atrium

Cardioneuroablation The procedure is performed under mild sedation (midazolam and fentanyl) using a 3.5 mm irrigated tip catheter (Navistar ThermoCool SmartTouch; Biosense Webster, Diamond Bar, California, USA) with contact force module and electroanatomical system Carto 3 (Biosense Webster, Diamond Bar, California, USA). After gaining transseptal access, an electroanatomical map of the right (RA) and left (LA) atrium is created and anatomically-based ablation of GP is performed. Ablation in the RA is started from the supero-posterior area (superior right atrial GP), to the middle-posterior area (posterior right atrial GP). In the LA, ablation is started at the site of the anterior right GP and is continued downwards along the anterior part of a common vestibulum of the right pulmonary veins (PV), opposite to the right-sided ablation lesions. Finally, area of right inferior GP, close to the RIPV is ablated under intracardiac echocardiography control. Using this technique, GP's located close to the left PV are not ablated. We use a pure anatomic approach without identification of GP by high-frequency stimulation or other imaging techniques.

Measurements.

1. Before CNA:

   1. Detailed history taking and assessment of eligibility
   2. Baseline 12-lead ECG for heart rate assessment, morphology and duration of the P wave and PR interval
   3. 24-hour Holter ECG for heart rhythm (mean, minimal, maximal, pauses) and heart rate variability (HRV) assessment
   4. Passive tilt test (70 degrees, 45 minutes) to fulfill inclusion criterion and to assess baseline autonomic parameters such as HRV and baroreflex sensitivity (BRS) using sequential method. These parameters will be calculated from 5 min recordings before and after orthostatic stress (tilt).
   5. Atropine test - positive response to intravenous atropine in a dose of 2 mg defined as at least 30% increase in sinus rate compared with baseline value
   6. Assessment of quality of life using the SF-36 questionnaire
   7. Implantable Loop Recorder (ILR) implantation 2-3 days before CNA
2. During CNA:

   1. Heart rate before and immediately after CNA
   2. Episodes of bradycardia (sinus arrest or atrio-ventrocular block) during application of RF to GP.
   3. Standard electrophysiological parameters (sinus node recovery time, corrected sinus recovery time, refractory atrio-ventricular node, atrio-ventricular conduction - Wenckebach point, A-H and H-V intervals) will be assessed before an immediately after CNA
   4. Atropine test (2 mg) will be repeated immediately after CNA.
3. After CNA:

   1. 1-2 days after CNA standard ECG
   2. Follow-up: 3, 12 and 24 months after CNA assessment of symptoms, 12 lead standard ECG, control ILR, 24-hour Holter ECG, tilt test and atropine test will be performed. Additionally, quality of life will be assessed using SF-36 questionnaire

      Definitions used for CNA efficacy assessment:
      * Complete efficacy - no syncope or presyncope during two years of follow-up
      * Partial efficacy - reduction of the number of syncopal (or presyncopal) episodes or change from syncopal to presyncopal episodes

      Primary endpoint

      - Time to first syncope recurrence

      Secondary endpoints
      * Syncope burden (number of syncopal episodes during two years)
      * Presyncope burden (number of presyncopal episodes during two years)
      * ILR: assessed heart rate and atrio-ventricular conduction if syncope occurs
      * CNA-induced changes in autonomic parameters
      * Prognostic value of autonomic parameters.
      * Safety of CNA: tamponade, stroke, phrenic nerve injury, permanent sinus arrest, local bleeding or vascular complications related to vascular access (hematoma / arteriovenous fistula)

      Statistical analysis Results will be presented as mean ± SD or numbers and percentages. Also CNA-induced changes(∆) in analysed parameters will be calculated. The ECG, electrophysiological and autonomic parameters obtained before and after CNA will be compared using student t-test or Mann-Whitney test where appropriate. The values of analysed parameters in predicting CNA efficacy will be assessed by computing sensitivity, specificity, positive and negative predictive value. The ROC curves will be drawn in order to establish optimal cut-off points of analysed parameters in predicting CNA efficacy.

      Anticipated results.

   <!-- -->

   1. CNA performed with technique used in the present study is effective in > 90% of patients.
   2. CNA-induced changes in analysed ECG and autonomic parameters predict CNA efficacy

ELIGIBILITY:
Inclusion Criteria:

* At least one documented spontaneous VVS during preceding 12 months or one syncope in history leading to injury and minimum 2 presyncopal events during preceding 12 months, refractory to all recommended types of standard treatment.
* In case of lack of ECG documentation during spontaneous syncope and history suggesting reflex syncope, at least 3 seconds of asystole due to sinus arrest or atrio-ventricular block with syncope or bradycardia <40 beats per minute with syncope or presyncope during baseline tilt test
* Sinus rhythm during ECG and tilt test
* Significantly decreased quality of life due to syncope
* Positive response to atropine test
* Obtained written informed consent.

Exclusion Criteria:

* Other possible and treatable causes of syncope such as significant cardiac disease, cardiac arrhythmia or abnormalities of vertebro-basiliar arteries
* History of stroke or TIA
* History of cardiac surgery
* Contraindications to ablation in the right or left atrium

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Time to first syncope recurrence. | Two-year follow-up after starting treatment.
  Recurrence of syncope (in days) after using the appropriate method (cardioneuroablation or standard non-pharmacological treatment).

SECONDARY OUTCOMES:
Syncope burden. | Two-year follow-up after starting treatment.
  Number of syncopal episodes (number of events during two-year follow-up).
Presyncope burden. | Two-year follow-up.
  Number of presyncopal episodes (number of events during two-year follow-up).
Heart rate and atrio-ventricular conduction if syncope occurs. | Two-year follow-up.
  Heart rate (beats/min) and longest pause (seconds) (based on ILR monitoring during syncope).
Cardioneuroablation-induced changes in heart rate variability predicting ablation efficacy. | 3, 12 and 24 months after cardioneuroablation.
  Cardioneuroablation-induced changes in heart rate variability (SDNN in msec) will be analyzed as a predictor of ablation efficacy.
Cardioneuroablation-induced changes in baroreflex sensitivity predicting ablation efficacy. | Two-year follow-up.
  Cardioneuroablation-induced changes in baroreflex sensitivity (msec/mmHg) will be analyzed as a predictor of ablation efficacy.
Complications associated with CNA procedure | Two-year follow-up.
  Assessment of possible complications: tamponade, stroke, phrenic nerve injury,(permanent sinus arrest, local bleeding or vascular complications related to vascular access (hematoma / arteriovenous fistula) - number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kulakowski, Prof., Study Chair — Centre of Postgraduate Medical Education; Roman Piotrowski, MD, PhD, Study Chair — Centre of Postgraduate Medical Education
Locations (1):
- Department of Cardiology, Postgraduate Medical School, Grochowski Hospital, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):1883-1948. doi: 10.1093/eurheartj/ehy037. No abstract available. PMID 29562304
- [Result] Grubb BP. Clinical practice. Neurocardiogenic syncope. N Engl J Med. 2005 Mar 10;352(10):1004-10. doi: 10.1056/NEJMcp042601. No abstract available. PMID 15758011
- [Result] Mathias CJ, Deguchi K, Schatz I. Observations on recurrent syncope and presyncope in 641 patients. Lancet. 2001 Feb 3;357(9253):348-53. doi: 10.1016/S0140-6736(00)03642-4. PMID 11210997
- [Result] Sheldon RS, Grubb BP 2nd, Olshansky B, Shen WK, Calkins H, Brignole M, Raj SR, Krahn AD, Morillo CA, Stewart JM, Sutton R, Sandroni P, Friday KJ, Hachul DT, Cohen MI, Lau DH, Mayuga KA, Moak JP, Sandhu RK, Kanjwal K. 2015 heart rhythm society expert consensus statement on the diagnosis and treatment of postural tachycardia syndrome, inappropriate sinus tachycardia, and vasovagal syncope. Heart Rhythm. 2015 Jun;12(6):e41-63. doi: 10.1016/j.hrthm.2015.03.029. Epub 2015 May 14. No abstract available. PMID 25980576
- [Result] Rose MS, Koshman ML, Spreng S, Sheldon R. The relationship between health-related quality of life and frequency of spells in patients with syncope. J Clin Epidemiol. 2000 Dec;53(12):1209-16. doi: 10.1016/s0895-4356(00)00257-2. PMID 11146266
- [Result] Bartoletti A, Fabiani P, Bagnoli L, Cappelletti C, Cappellini M, Nappini G, Gianni R, Lavacchi A, Santoro GM. Physical injuries caused by a transient loss of consciousness: main clinical characteristics of patients and diagnostic contribution of carotid sinus massage. Eur Heart J. 2008 Mar;29(5):618-24. doi: 10.1093/eurheartj/ehm563. Epub 2007 Dec 16. PMID 18086659
- [Result] Chen-Scarabelli C, Scarabelli TM. Neurocardiogenic syncope. BMJ. 2004 Aug 7;329(7461):336-41. doi: 10.1136/bmj.329.7461.336. No abstract available. PMID 15297344
- [Result] Brignole M, Menozzi C, Moya A, Andresen D, Blanc JJ, Krahn AD, Wieling W, Beiras X, Deharo JC, Russo V, Tomaino M, Sutton R; International Study on Syncope of Uncertain Etiology 3 (ISSUE-3) Investigators. Pacemaker therapy in patients with neurally mediated syncope and documented asystole: Third International Study on Syncope of Uncertain Etiology (ISSUE-3): a randomized trial. Circulation. 2012 May 29;125(21):2566-71. doi: 10.1161/CIRCULATIONAHA.111.082313. Epub 2012 May 7. PMID 22565936
- [Result] Aydin MA, Mortensen K, Salukhe TV, Wilke I, Ortak M, Drewitz I, Hoffmann B, Mullerleile K, Sultan A, Servatius H, Steven D, von Kodolitsch Y, Meinertz T, Ventura R, Willems S. A standardized education protocol significantly reduces traumatic injuries and syncope recurrence: an observational study in 316 patients with vasovagal syncope. Europace. 2012 Mar;14(3):410-5. doi: 10.1093/europace/eur341. Epub 2011 Nov 1. PMID 22048993
- [Result] Sheldon RS, Morillo CA, Klingenheben T, Krahn AD, Sheldon A, Rose MS. Age-dependent effect of beta-blockers in preventing vasovagal syncope. Circ Arrhythm Electrophysiol. 2012 Oct;5(5):920-6. doi: 10.1161/CIRCEP.112.974386. Epub 2012 Sep 12. PMID 22972872
- [Result] Tan MP, Newton JL, Chadwick TJ, Gray JC, Nath S, Parry SW. Home orthostatic training in vasovagal syncope modifies autonomic tone: results of a randomized, placebo-controlled pilot study. Europace. 2010 Feb;12(2):240-6. doi: 10.1093/europace/eup368. Epub 2009 Nov 17. PMID 19919966
- [Result] Romme JJ, van Dijk N, Go-Schon IK, Reitsma JB, Wieling W. Effectiveness of midodrine treatment in patients with recurrent vasovagal syncope not responding to non-pharmacological treatment (STAND-trial). Europace. 2011 Nov;13(11):1639-47. doi: 10.1093/europace/eur200. Epub 2011 Jul 13. PMID 21752826
- [Result] Raviele A, Giada F, Menozzi C, Speca G, Orazi S, Gasparini G, Sutton R, Brignole M; Vasovagal Syncope and Pacing Trial Investigators. A randomized, double-blind, placebo-controlled study of permanent cardiac pacing for the treatment of recurrent tilt-induced vasovagal syncope. The vasovagal syncope and pacing trial (SYNPACE). Eur Heart J. 2004 Oct;25(19):1741-8. doi: 10.1016/j.ehj.2004.06.031. PMID 15451153
- [Result] Yao Y, Shi R, Wong T, Zheng L, Chen W, Yang L, Huang W, Bao J, Zhang S. Endocardial autonomic denervation of the left atrium to treat vasovagal syncope: an early experience in humans. Circ Arrhythm Electrophysiol. 2012 Apr;5(2):279-86. doi: 10.1161/CIRCEP.111.966465. Epub 2012 Jan 24. PMID 22275485
- [Result] Pachon JC, Pachon EI, Cunha Pachon MZ, Lobo TJ, Pachon JC, Santillana TG. Catheter ablation of severe neurally meditated reflex (neurocardiogenic or vasovagal) syncope: cardioneuroablation long-term results. Europace. 2011 Sep;13(9):1231-42. doi: 10.1093/europace/eur163. Epub 2011 Jun 28. PMID 21712276
- [Result] Aksu T, Golcuk E, Yalin K, Guler TE, Erden I. Simplified Cardioneuroablation in the Treatment of Reflex Syncope, Functional AV Block, and Sinus Node Dysfunction. Pacing Clin Electrophysiol. 2016 Jan;39(1):42-53. doi: 10.1111/pace.12756. Epub 2015 Oct 26. PMID 26411271
- [Result] Sun W, Zheng L, Qiao Y, Shi R, Hou B, Wu L, Guo J, Zhang S, Yao Y. Catheter Ablation as a Treatment for Vasovagal Syncope: Long-Term Outcome of Endocardial Autonomic Modification of the Left Atrium. J Am Heart Assoc. 2016 Jul 8;5(7):e003471. doi: 10.1161/JAHA.116.003471. PMID 27402231
- [Result] Piotrowski R, Baran J, Kulakowski P. Cardioneuroablation using an anatomical approach: a new and promising method for the treatment of cardioinhibitory neurocardiogenic syncope. Kardiol Pol. 2018;76(12):1736-1738. doi: 10.5603/KP.a2018.0200. Epub 2018 Oct 19. No abstract available. PMID 30338504
- [Derived] Piotrowski R, Baran J, Sikorska A, Krynski T, Kulakowski P. Cardioneuroablation for Reflex Syncope: Efficacy and Effects on Autonomic Cardiac Regulation-A Prospective Randomized Trial. JACC Clin Electrophysiol. 2023 Jan;9(1):85-95. doi: 10.1016/j.jacep.2022.08.011. Epub 2022 Aug 28. PMID 36114133